CLINICAL TRIAL: NCT07394816
Title: The Effect of Ultrasound-Guided Fascial Plane Blocks on Postoperative Pulmonary Complications in Patients Undergoing Major Abdominal Surgery: A Prospective Observational Study
Brief Title: Can Ultrasound-Guided Fascial Plane Blocks Reduce Postoperative Pulmonary Complications After Major Abdominal Surgery?
Acronym: FPB-PPC
Status: Not yet recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arif Timuroğlu, MD, Specialist in Anesthesiology and Intensive Care, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-12/186
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pulmonary Complications (PPCs); Abdominal Surgeries; Postoperative Pain Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fascial Plane Block Group: Patients undergoing elective major abdominal surgery who receive an ultrasound-guided fascial plane block at the end of surgery as part of routine clinical practice for postoperative analgesia. The decision to perform the block is made by the responsible anesthesia team and is not influenced by the study protocol.
- Control Group: Patients undergoing elective major abdominal surgery who do not receive an ultrasound-guided fascial plane block and are managed with other routine postoperative analgesic methods, including epidural analgesia, intravenous patient-controlled analgesia, or oral analgesics, according to standard clinical practice.

SUMMARY:
This prospective observational study aims to evaluate whether the use of ultrasound-guided fascial plane blocks is associated with a lower incidence of postoperative pulmonary complications in adult patients undergoing elective major abdominal surgery under general anesthesia.

Patients will be observed in two groups based on routine clinical practice: those who receive an ultrasound-guided fascial plane block for postoperative analgesia and those managed with other standard analgesic methods. The choice of analgesic technique will be determined by the responsible anesthesia team and not influenced by the study.

Postoperative pulmonary complications occurring within the first 7 days after surgery will be recorded using reopening the European Perioperative Clinical Outcome (EPCO) criteria. Secondary outcomes will include unplanned intensive care unit admission, length of hospital stay, and 30-day mortality. No additional procedures or interventions will be performed for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Scheduled for elective major abdominal surgery (e.g., colorectal, hepatobiliary, pancreatic, or gastric surgery)
* ASA physical status II-III
* Ability to provide written informed consent
* Planned use of general anesthesia with or without adjunct regional techniques

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Known allergy or contraindication to local anesthetics
* Coagulopathy or ongoing anticoagulant therapy contraindicating regional anesthesia
* Infection at the site of planned block
* Pre-existing chronic opioid use or chronic pain syndrome
* Severe hepatic, renal, or cardiac failure (e.g., Child-Pugh C, end-stage renal disease, EF <30%)
* Cognitive impairment or severe dementia preventing adequate pain assessment
* Emergency surgery
* Body mass index (BMI > 40 kg/m²)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of patients aged 65 years and older who are scheduled to undergo elective major abdominal surgery under general anesthesia. Eligible participants will be managed in a tertiary care hospital and will be allocated to either a fascial plane block group or a control group receiving standard perioperative analgesia. The study aims to evaluate postoperative outcomes in an elderly surgical population with comparable baseline characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications (PPCs) | Within the first 7 postoperative days
  Postoperative pulmonary complications will be defined and recorded according to the European Perioperative Clinical Outcome (EPCO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: arif timuroglu, Principal Investigator — Dr. Abdurrahman yurtaslan Ankara Oncology Hospital
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Hospital, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies and concerns regarding patient confidentiality and data protection.